CLINICAL TRIAL: NCT02316561
Title: Single Dose Ablative Preoperative Radiation Treatment for Early-Stage Breast Cancer in Elderly Patients
Brief Title: Single Dose Ablative Radiation Treatment for Early-Stage Breast Cancer
Acronym: ABLATIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, K.R. Charaghvandi, MD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL46017.041.13
Record Dates: First submitted 2014-10-10; First posted 2014-12-15 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single dose ablative radiotherapy (Experimental): Eligible patients for single dose ablative radiotherapy according to inclusion and exclusion criteria
  Interventions: Radiation: Single dose ablative radiotherapy

INTERVENTIONS:
Radiation: Single dose ablative radiotherapy — A single dose ablative radiotherapy will be delivered prior to surgery

SUMMARY:
The purpose of the study is to investigate the feasibility of a preoperative, single dose, ablative partial breast radiation treatment in patients with early-stage breast cancer.

DETAILED DESCRIPTION:
A total of twenty-five patients will be treated with a single dose preoperative ablative radiation treatment. After a vigilant follow-up with MRI, breast conserving surgery will be performed 6 months after the ablative radiation treatment. The total follow-up time is 10 years.

This study aims to present an ablative radiotherapy treatment approach that could resolve to some extent the disadvantages of current breast conserving treatment in elderly low-risk breast cancer patients who are currently not treated according to guidelines due to co-morbidity.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance scale ≤2.
* Females at least 50 years of age with unifocal cT1N0 breast cancer or females at least 70 years of age with an unifocal cT1-2(maximum 3 cm)N0 breast cancer:

  - Tumor size as assessed on MRI
* On tumor biopsy:

  * Non-lobular invasive histological type carcinoma.
  * LCIS is accepted.
  * ER positive tumor receptor.
* Tumor negative sentinel node.
* Adequate communication and understanding skills of the Dutch language.

Exclusion Criteria:

* Legal incapacity
* Indication for chemotherapy or immunotherapy (i.e. patients with an indication for endocrine therapy are eligible)
* BRCA gene mutation.
* Previous history of breast cancer
* Other type of malignancy within 5 years before breast cancer diagnosis. For adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin no specific time span from breast cancer diagnosis is required for inclusion
* Her2neu positive tumor.
* Previous history of ipsilateral breast surgery and impaired cosmetic outcome, as assessed by the treating surgeon or radiation-oncologist.
* Collagen synthesis disease.
* Signs of extensive DCIS component on histological biopsy or mammogram.
* Invasive lobular carcinoma.
* MRI absolute contraindications as defined by the Radiology Department.
* Nodal involvement with cytological or histological confirmation.
* Treatment with neo-adjuvant systemic therapy.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Pathological complete response | 6 months after radiotherapy

SECONDARY OUTCOMES:
Radiological tumor response on MRI according to the RECIST criteria | Within 1 week and 2, 4 and 6 months after radiotherapy
Radiological tumor response on FDG-PET-CT according to the PERCIST criteria | At 6 months after radiotherapy
Quality of life according to EORTC QLQ-BR23 and EORTC QLQ-C30 questionnaires | Until 10 years after radiotherapy
Cosmetic results as assessed by patient questionnaire, radiation oncologist evaluation and BCCT.core software | Until 10 years after radiotherapy
Frailty assessment according to the Groningen Frailty Indicator | Until 10 years after radiotherapy
Functionality assessment using patient questionnaires on physical activity and the Hospital Anxiety and Depression Scale questionnaire. | Until 10 years after radiotherapy
Local relapse rates | Until 10 years after radiotherapy
Regional relapse rates | Until 10 years after radiotherapy
Distant relapse rates | Until 10 years after radiotherapy
Disease free survival | Until 10 years after radiotherapy
Overall survival | Until 10 years after radiotherapy

OTHER OUTCOMES:
Tumor related genetic characteristics associated with radiotherapy responsiveness | Until 10 years after radiotherapy
  Future research proposal performed within 10 years after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: HJGD van den Bongard, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groot Koerkamp ML, de Hond YJM, Maspero M, Kontaxis C, Mandija S, Vasmel JE, Charaghvandi RK, Philippens MEP, van Asselen B, van den Bongard HJGD, Hackett SS, Houweling AC. Synthetic CT for single-fraction neoadjuvant partial breast irradiation on an MRI-linac. Phys Med Biol. 2021 Apr 16;66(8). doi: 10.1088/1361-6560/abf1ba. PMID 33761491
- [Derived] Charaghvandi RK, van Asselen B, Philippens ME, Verkooijen HM, van Gils CH, van Diest PJ, Pijnappel RM, Hobbelink MG, Witkamp AJ, van Dalen T, van der Wall E, van Heijst TC, Koelemij R, van Vulpen M, van den Bongard HJ. Redefining radiotherapy for early-stage breast cancer with single dose ablative treatment: a study protocol. BMC Cancer. 2017 Mar 9;17(1):181. doi: 10.1186/s12885-017-3144-5. PMID 28274211